CLINICAL TRIAL: NCT01026194
Title: A Phase III Study of MP-513 in Combination With Thiazolidinedione in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of MP-513 in Combination With Thiazolidinedione in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A7
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Pemoline; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo / Teneli + Pio (Placebo Comparator)
  Interventions: Drug: Placebo / Teneli (Teneligliptin) + pio (pioglitazone)
- Teneli / Teneli + pio (Experimental)
  Interventions: Drug: Teneli / Teneli + pio

INTERVENTIONS:
Drug: Placebo / Teneli (Teneligliptin) + pio (pioglitazone) — Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone.
  Arms: Placebo / Teneli + Pio
Drug: Teneli / Teneli + pio — Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone.
  Arms: Teneli / Teneli + pio

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MP-513 (Teneligliptin) in combination with thiazolidinedione (pioglitazone) in patients with type 2 Diabetes for 12 weeks administration and to evaluate the safety and efficacy of MP-513 in combination with thiazolidinedione with an extension treatment for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 - 75 years old
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is between 6.5% and 10.0%
* Patients who took Thiazolidinedione for diabetes over 16 weeks before administration of investigational drug
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients who are accepting treatments of arrhythmias
* Patients with serious diabetic complications
* Patients who are the excessive alcohol addicts
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Shinjukuku, Tokyo, Japan

REFERENCES:
- [Derived] Kadowaki T, Kondo K. Efficacy and safety of teneligliptin in combination with pioglitazone in Japanese patients with type 2 diabetes mellitus. J Diabetes Investig. 2013 Nov 27;4(6):576-84. doi: 10.1111/jdi.12092. Epub 2013 May 27. PMID 24843712
- [Derived] Kadowaki T, Kondo K. Efficacy and safety of teneligliptin added to glimepiride in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled study with an open-label, long-term extension. Diabetes Obes Metab. 2014 May;16(5):418-25. doi: 10.1111/dom.12235. Epub 2013 Dec 10. PMID 24205974

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Teneli + Pio: Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone.
- Teneli/Teneli + Pio: Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone.
Period: Period 1：Double Blind Period
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Started | 101 | 103
Completed | 98 | 98
Not Completed | 3 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 4
Period: Period 2：Open-label Period
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Started | 98 | 98
Completed | 91 | 88
Not Completed | 7 | 10
Not completed — Adverse Event | 4 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.9) | 59.7 (9.7) | 60.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 35 | 60
  Male | 76 | 68 | 144

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate.
Time Frame: at Week 0 and Week 12
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization. Analysis based on last observation carried forward, where the last postbaseline double-blind observed value was carried forward and used for Week 12 where data was missing.
Measure: Least Squares Mean (Standard Error); unit: Percent of HbA1c
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Number analyzed (Participants) | 101 | 103
Percent of HbA1c | -0.20 (0.05) | -0.94 (0.04)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: The change from Baseline in Fasting Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline Fasting Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Number analyzed (Participants) | 101 | 103
mg / dL | -4.5 (2.0) | -21.0 (1.9)

3. Secondary Outcome: Change From Baseline in the Areas Under the Curve From 0 to 2 h (AUC0-2h) for Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in AUC0-2h for Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline AUC0-2h for Postprandial Plasma Glucose as a covariate.
Time Frame: 0, 0.5, 1, 2 hours post-dose at Week 0 and Week 12
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization.
Measure: Least Squares Mean (Standard Error); unit: mg*h / dL
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Number analyzed (Participants) | 98 | 98
mg*h / dL | -13.722 (5.134) | -85.031 (5.134)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in 2-hour Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline 2-hour Postprandial Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo/Teneli + Pio | Teneli/Teneli + Pio
Number analyzed (Participants) | 98 | 98
mg / dL | -5.6 (3.6) | -56.9 (3.6)

ADVERSE EVENTS:
Groups:
- Placebo/Teneli + Pio (Data Through Week 12): Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone. The adverse events which occured from Week 0 to Week 12 were shown.
- Teneli/Teneli + Pio (Data Through Week 12): Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone. The adverse events which occured from Week 0 to Week 12 were shown.
- Placebo/Teneli + Pio (Data From Week 12 to Week 52): Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone. The adverse events which occured from Week 12 to Week 52 were shown.
- Teneli/Teneli + Pio (Data Through Week 52): Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with pioglitazone. The adverse events which occured from Week 12 to Week 52 were shown.
Arm/Group | Placebo/Teneli + Pio (Data Through Week 12) | Teneli/Teneli + Pio (Data Through Week 12) | Placebo/Teneli + Pio (Data From Week 12 to Week 52) | Teneli/Teneli + Pio (Data Through Week 52)
Serious Adverse Events (participants affected / at risk) | 1/101 | 4/103 | 3/98 | 11/103
Other Adverse Events (participants affected / at risk) | 47/101 | 63/103 | 89/98 | 88/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli + Pio (Data Through Week 12) (N=101) | Teneli/Teneli + Pio (Data Through Week 12) (N=103) | Placebo/Teneli + Pio (Data From Week 12 to Week 52) (N=98) | Teneli/Teneli + Pio (Data Through Week 52) (N=103)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli + Pio (Data Through Week 12) (N=101) | Teneli/Teneli + Pio (Data Through Week 12) (N=103) | Placebo/Teneli + Pio (Data From Week 12 to Week 52) (N=98) | Teneli/Teneli + Pio (Data Through Week 52) (N=103)
Abscess (Infections and infestations) | 0 | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 4 | 2
Cystitis (Infections and infestations) | 3 | 1 | 2 | 4
Nasal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 12 | 33 | 33
Pharyngitis (Infections and infestations) | 0 | 1 | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 2
Gastritis viral (Infections and infestations) | 0 | 1 | 0 | 1
Herpes dermatitis (Infections and infestations) | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 2 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 3 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 2
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 2 | 3
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 4 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 4 | 3
Headache (Nervous system disorders) | 1 | 2 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 3 | 2
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 1 | 1
Spinocerebellar disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrovascular stenosis (Nervous system disorders) | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 2 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 2 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 2
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 2 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 10 | 11
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 4 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 1 | 4
Gastritis (Gastrointestinal disorders) | 0 | 2 | 4 | 6
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 2 | 4 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric xanthoma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Supernumerary teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 6
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6 | 7
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Calculus prostatic (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 2 | 0
Oedema peripheral (General disorders) | 6 | 2 | 4 | 4
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 4 | 9
Blood triglycerides increased (Investigations) | 1 | 2 | 1 | 5
Blood urea increased (Investigations) | 1 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1
Glucose urine present (Investigations) | 8 | 3 | 6 | 7
Blood urine present (Investigations) | 2 | 3 | 5 | 12
White blood cell count increased (Investigations) | 0 | 1 | 2 | 1
Protein urine present (Investigations) | 1 | 4 | 3 | 9
Urine ketone body present (Investigations) | 2 | 0 | 6 | 2
Occult blood positive (Investigations) | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 5
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 4
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other